CLINICAL TRIAL: NCT02256059
Title: Treatment of Displaced Lateral Clavicle Fractures Using a Locking Compression Plate With Lateral Extension - Clinical Observational Study
Brief Title: Treatment of Displaced Lateral Clavicle Fractures Using a Locking Compression Plate With Lateral Extension
Acronym: LatClav
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, MD, Technical University of Munich
Other Study IDs: Beiromat_03
Record Dates: First submitted 2014-09-28; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Fracture, Closed, Comminuted, Healing
MeSH Terms: conditions — Fractures, Bone; Fractures, Comminuted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plate osteosynthesis: Patients with fracture of the lateral clavicle and indication for surgical treatment
  Interventions: Procedure: Plate osteosynthesis

INTERVENTIONS:
Procedure: Plate osteosynthesis — Plate osteosynthesis using LCP plate (Synthes)

SUMMARY:
Treatment of lateral fractures of the clavicle is challenging and has been controversially discussed for a long time due to high non-union rates in non-operative treatment and high complication rates in surgical treatment. A recently developed implant was proven to ensure a biomechanically sufficient fixation of fractures leading to bony union and promising functional outcome in a small collective of patients.

DETAILED DESCRIPTION:
Treatment of lateral fractures of the clavicle is challenging and has been controversially discussed for a long time due to high non-union rates in non-operative treatment and high complication rates in surgical treatment. A recently developed implant was proven to ensure a biomechanically sufficient fixation of fractures leading to bony union and promising functional outcome in a small collective of patients.

In this prospective study patients with dislocated fractures of the lateral clavicle (Jäger&Breitner I-III, Neer I-III) are enrolled. All patients are surgically treated using the locking compression plate (LCP) for the superior anterior clavicle (Synthes®). Functional outcome is recorded using the Munich Shoulder Questionnaire (MSQ) allowing for qualitative self-assessment of the Shoulder Pain and Disability Index (SPADI), of the Disability of the Arm, Shoulder and Hand (DASH) score and of the Constant Score. Acromioclavicular joint stability is evaluated using the Taft-Score.

ELIGIBILITY:
Inclusion Criteria:

* Dislocated fracture of the lateral clavicle
* Informed consent.

Exclusion Criteria:

* Patients with a history of any other pathology such as preexisting rotator cuff tear, gleno-humeral instability, glenohumeral osteoarthritis (> Samilson I), Acromioclavicular joint instability, Acromioclavicular osteoarthritis, calcifying tendonitis, biceps pathology or signs of cervical root symptoms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from a dislocated fracture of the lateral clavicle presenting at our emergency department.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
bone healing | 12 month
  time until bone healing, visualized using conventional x-ray in two planes

SECONDARY OUTCOMES:
shoulder function | 12 month
  shoulder function assessed using Munich Shoulder Questionnaire [MSQ]

CONTACTS AND LOCATIONS:
Overall Officials: Chlodwig Kirchhoff, MD, Principal Investigator — Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Technische Universität München
Locations (1):
- Klinik und Poliklinik für Unfallchirurgie, Klinikum rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Beirer M, Siebenlist S, Cronlein M, Postl L, Huber-Wagner S, Biberthaler P, Kirchhoff C. Clinical and radiological outcome following treatment of displaced lateral clavicle fractures using a locking compression plate with lateral extension: a prospective study. BMC Musculoskelet Disord. 2014 Nov 19;15:380. doi: 10.1186/1471-2474-15-380. PMID 25406639